CLINICAL TRIAL: NCT05250908
Title: A Prospective, Randomized Clinical Trial Evaluating INTIBIA, an Investigational Implantable Tibial Nerve Stimulator, Through 24-Months (INTIBIA Pivotal Study IU024)
Brief Title: INTIBIA Pivotal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IU024
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence, Urge; Urinary Bladder, Overactive; Urinary Bladder Diseases; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Manifestations
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive; Urinary Bladder Diseases; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Manifestations

STUDY DESIGN:
Intervention Model Description: All eligible subjects will be implanted with the INTIBIA device. Subjects will be randomized to either INTIBIA therapeutic or INTIBIA non-therapeutic in a 2:1 ratio for the first 3 months of the study, at which point all subjects will receive therapeutic stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects and investigator/site personnel are blinded until the Month 3 visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- INTIBIA Therapeutic (Experimental): Implanted with INTIBIA device and programmed to therapeutic stimulation for the duration of the study.
  Interventions: Device: INTIBIA Therapeutic
- INTIBIA Non-Therapeutic (Experimental): Implanted with INTIBIA device and programmed to non-therapeutic stimulation for the first 3 months, then to therapeutic stimulation for the duration of the study.
  Interventions: Device: INTIBIA Non-Therapeutic

INTERVENTIONS:
Device: INTIBIA Therapeutic — INTIBIA implantable tibial nerve stimulator with therapeutic stimulation
  Arms: INTIBIA Therapeutic
Device: INTIBIA Non-Therapeutic — INTIBIA implantable tibial nerve stimulator with non-therapeutic stimulation for 3 months, then therapeutic stimulation
  Arms: INTIBIA Non-Therapeutic

SUMMARY:
Prospective, randomized, double-blind, multicenter study to evaluate the safety and efficacy of an implantable tibial nerve stimulator in subjects with urgency urinary incontinence (UUI).

DETAILED DESCRIPTION:
All eligible subjects will be implanted with the INTIBIA device. Subjects will be randomized to either INTIBIA therapeutic or INTIBIA non-therapeutic in a 2:1 ratio for the first 3 months of the study, at which point all subjects will receive therapeutic stimulation. Subjects will complete voiding diaries and questionnaires at Baseline and prior to each follow-up visit, which will occur at Months 3, 6, 12, and 24. Subjects will be offered to keep the device or have it explanted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women or men 22-80 years of age
* Symptoms of overactive bladder with urgency urinary incontinence (UUI) demonstrated on a 72-hour voiding diary defined as a minimum of four (4) leaking episodes associated with urgency, and at least one leaking episode each 24-hour period
* Greater than or equal to 6-month history of UUI diagnosis
* Failure of conservative or behavioral therapy (e.g., bladder diet, timed voiding, bladder training, bladder control strategies, pelvic floor muscle training, fluid management)
* Willing to abstain from OAB medications for the duration of the study
* Willing to maintain a stable dose of all other medications that affect bladder function (e.g., tricyclic antidepressants) for at least four (4) weeks prior to beginning the baseline voiding diary and baseline questionnaires
* Ambulatory and able to use the toilet independently and without difficulty
* Willing and capable of providing informed consent
* Willing and able to complete all procedures and follow-up visits indicated in the protocol

Exclusion Criteria:

* Diagnosis of stress urinary incontinence or mixed urinary incontinence, as confirmed by cough stress test and with a response of Yes to Q3 on the UDI-6 questionnaire
* Current symptomatic urinary tract infection (UTI), urethritis, or more than three (3) UTIs in past year
* Have post-void residual urine volume >30% of total voided volume
* Inadequate skin integrity, any evidence of an infection, or lower leg edema limiting placement of device per physician discretion
* Evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject
* Prior treatment of urinary symptoms with nerve stimulation (e.g., percutaneous tibial nerve stimulation [PTNS] or sacral nerve stimulation [SNS])
* History of chronic pain (e.g., chronic pelvic pain, fibromyalgia, Lyme disease, chronic back pain)
* An active implantable electronic device regardless of whether stimulation is ON or OFF
* Treatment of urinary symptoms with botulinum toxin therapy within six (6) months
* Any neurological condition that could interfere with normal bladder or tibial nerve function, including debilitating stroke, epilepsy, multiple sclerosis, Parkinson's disease, peripheral neuropathy, fibromyalgia, or spinal cord injury (e.g., paraplegia)
* Current urinary tract mechanical obstruction (e.g., benign prostatic enlargement or urethral stricture)
* Other urinary tract dysfunction (e.g., abnormal upper urinary tract function, vesicoureteral reflux, bladder stone or tumor, urinary fistula)
* End stage renal failure, GFR < 35, or dialysis
* History of pelvic cancer requiring radiation or chemotherapy treatment within the past two years
* Pelvic organ prolapse at or beyond the hymenal ring
* Interstitial cystitis or bladder pain syndrome as defined by either American Urological Association (AUA) or European Association of Urology (EAU) guidelines prior to INTIBIA implant date
* Diabetes with peripheral nerve compromise or uncontrolled diabetes
* Pregnant as confirmed by urine or serum pregnancy test, plans to become pregnant over the study period, is less than one-year post-partum, is breast-feeding
* Current active or a chronic systemic infection
* Condition requiring magnetic resonance imaging (MRI) of lower leg
* Condition requiring diathermy
* Allergy to polyethylene terephthalate, silicone rubber, platinum, iridium, or polyurethane
* Allergy to local anesthetic or adhesives
* Deemed unsuitable for enrollment by the investigator based on history or physical examination (e.g., bleeding disorders, current anticoagulant medications)
* Enrolled in another investigational or interventional device or drug trial over the study period

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 3 Months
  ≥50% reduction in UUI episodes between INTIBIA therapeutic and INTIBIA non-therapeutic
Response Rate | 12 Months
  ≥50% reduction in UUUI episodes in the INTIBIA therapeutic group

SECONDARY OUTCOMES:
Urgency Score | 3 Months
  Change in mean urgency score relative to baseline on a scale of 0 (no urgency) to 4 (urge incontinence)
Daily Voids | 3 Months
  Change in mean number of daily voids relative to baseline

OTHER OUTCOMES:
Response Rate | 6 Months
  ≥50% reduction in UUUI episodes in the INTIBIA therapeutic group
Response Rate | 3, 6, and 12 Months
  ≥50% reduction in number of voids or a return to normal voiding frequency (< 8 voids/day)
Daily Voids | 6 and 12 Months
  Change in mean number of daily voids relative to baseline
Urgency Score | 6 and 12 Months
  Change in mean urgency score relative to baseline on a scale of 0 (no urgency) to 4 (urge incontinence)
International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form | 3, 6, and 12 Months
  Change in ICIQ-UI SF questionnaire total score compared to baseline. Scoring 0 (best outcome) - 21 (worst outcome)
OverActive Bladder questionnaire - Short Form | 3, 6, and 12 Months
  Change in the OABq-SF questionnaire total score compared to baseline. Scoring 1 (best) - 6 (worst) on 19 questions.
Dry | 3, 6, and 12 Months
  The proportion of dry subjects, defined as those with 0 incontinence episodes associated with urgency as captured on the 72-hour voiding diary
Patient's Global Impression of Improvement Questionnaire | 3, 6, and 12 Months
  The proportion of subjects reporting "much better" or "very much better" on the Patient Global Impression of Improvement (PGI-I) questionnaire
Surgical Satisfaction Questionnaire (SSQ-8) | 3 Months
  Surgical Satisfaction Questionnaire (SSQ-8)
EQ-5D-5L Questionnaire | 3, 6, and 12 Months
  Change in the EQ-5D-5L index score compared to baseline, on a 1-5 scale with 1 being the best outcome and 5 being the worst outcome. VAS scale measures overall health with 0 being the worst outcome and 100 being the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Principal Investigator — Wake Forest University
Locations (22):
- United States (20):
  - Cedars-Sinai Medical Group, Beverly Hills, California
  - Urology Group of Southern California, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advanced Urology Associates, Daytona Beach, Florida
  - Southeastern Urogynecology & Pelvic Surgery, Moultrie, Georgia
  - Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Advanced Urogynecology of Michigan, Dearborn, Michigan
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Atlantic Health System - AMG Urology (Garden State Urology), Denville, New Jersey
  - Wake Forest University, Winston-Salem, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - MetroHealth System, Cleveland, Ohio
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery- Axia Womens Health, Allentown, Pennsylvania
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - The Female Pelvic Health Center, Newtown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Houston Metro Urology, Houston, Texas
- Netherlands (2):
  - Bergman Clinics, Women's Health, Department of Gynecology, Amsterdam
  - Isala Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: No